CLINICAL TRIAL: NCT02720029
Title: Detection of Silent Aspiration Events Utilizing pH/Impedance Probes in Hospitalized Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with enrollment
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Joshua Fessel, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 141751
Record Dates: First submitted 2016-03-14; First posted 2016-03-25 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Acid Aspiration Syndrome
Keywords: aspiration; reflux
MeSH Terms: conditions — Pneumonia, Aspiration; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pH/impedance monitor (Experimental)
  Interventions: Device: pH/impedance monitor

INTERVENTIONS:
Device: pH/impedance monitor — Placement of pH/impedance monitor via the nasogastric route with monitoring for 24 hours, followed by removal.

SUMMARY:
Monitoring and quantification of reflux events in high risk critically ill inpatients and lower risk general medical/surgical inpatients, with comparison to relevant clinical variables.

DETAILED DESCRIPTION:
The investigators will conduct a pilot prospective cohort study of the incidence of reflux of gastric contents into the esophagus and the correlation with clinically evident aspiration events. The investigators will demonstrate that an esophageal multichannel pH/impedance probe can be used safely and effectively in an inpatient population to monitor reflux of acidic and non-acidic contents into the esophagus. The investigators will determine the frequency and severity of reflux events in a 24 hour period in two hospitalized patient populations: general medicine patients on the wards and critically ill patients in the intensive care unit. The investigators will then examine the relationship between the documented reflux events and clinically apparent aspiration events. The incidence of these silent reflux events in hospitalized patients is currently unclear.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Admitted to medical-surgical floor or medical intensive care unit

Exclusion Criteria:

1. Patients with contraindication to nasogastric tube placement (facial trauma, active epistaxis, abnormal nasopharyngeal or facial anatomy, esophageal stricture or injury, esophageal varices)
2. Patients requiring non-invasive positive pressure ventilation
3. Patients with uncontrolled vomiting
4. Patients with planned or anticipated airway or esophageal procedure within the 24-hour monitoring period
5. Patients not expected to survive for 24 hours or those receiving hospice/palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Number of reflux events | 24 hours
  Summation of acid reflux events and non-acid reflux events over 24hr monitoring period measured by pH change and impedance change detected by the probe

SECONDARY OUTCOMES:
Clinically apparent aspiration events | Duration of hospitalization, on average 14 days
  Counting clinically apparent aspiration events by way of manual chart review
Combined aspiration event endpoint | Duration of hospitalization, on average 14 days
  Summation of clinically apparent aspiration events, new infiltrates on chest imaging, increase in oxygen requirements, or need for higher level of care due to respiratory decompensation - all components determined by manual chart review

CONTACTS AND LOCATIONS:
Overall Officials: Joshua P Fessel, MD, PhD, Principal Investigator — Vanderbilt University

IPD SHARING:
Plan to Share IPD: Yes